CLINICAL TRIAL: NCT03925259
Title: A Pilot Randomised Dismantling Trial of the Efficacy of Self-As-Context During Acceptance and Commitment Therapy
Brief Title: Dismantling the Efficacy of Self-As-Context During Acceptance and Commitment Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Stephen Kellett, IAPT Programme Director, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 144363
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Depression, Anxiety
Keywords: ACT; dismantling; long term conditions
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: The design was a pilot, randomised and controlled dismantling trial. Ethical approval was granted to conduct the trial (ref: 144363) and was contingent on adverse events being monitored in the arms. Participants were randomised to either full-ACT (i.e. the full hexaflex approach) or ACT-SAC (i.e. ACT minus the self-as-context component of the hexaflex). Participants were blind to their allocation. ACT process measures were completed at assessment, final therapy session and at 6-week follow-up and the outcome measures were taken on a session-by-session basis and at 6-week follow-up.
Who Masked: Participant
Masking Description: The participants were masked as to their allocation to either full treatment or treatment with the self-as-context component removed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-ACT (Active Comparator): Participants received eight 50-minute sessions of ACT. A treatment protocol comprising of eight modules in the Full-ACT arm was developed by the research team. Each module comprised a series of exercises and metaphors, as well as guidance on how to discuss specific components. There was some degree of flexibility by which therapists introduced modules (Strosahl et al., 2004). However, by the final session, all eight mandatory subjects, exercises, and metaphors had to be covered. Modules were as follows: creative hopelessness; acceptance; defusion; present-momentness; self-as-context; values; and committed action.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- ACT-SAC (Experimental): Participants received eight 50-minute sessions of ACT. A treatment protocol comprising of seven modules in the ACT-SAC arm was developed by the research team. Each module comprised a series of exercises and metaphors, as well as guidance on how to discuss specific components. There was some degree of flexibility by which therapists introduced modules (Strosahl et al., 2004). However, by the final session, all mandatory subjects, exercises, and metaphors had to be covered. Modules were as follows: creative hopelessness; acceptance; defusion; present-momentness; values; and committed action.
  The ACT-SAC condition removed the self-as-context module; therapists were instructed to avoid any reference to self-as-context or to support discussions regarding this process.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and commitment therapy (ACT) is a 'third wave' behaviour therapy delivered on a one to one basis.

SUMMARY:
The six processes within the psychological flexibility model of acceptance and commitment therapy (ACT) are seen as being equally theoretically and clinically important. The utility of self-as-context component however has never been isolated in a dismantling study. The present study therefore sought to conduct a pilot two-arm dismantling component study of ACT, quarantining the self-as-context component from one of the arms. Patients with a long-term health condition (LTC) and concurrent mental health condition were randomised into one of two study arms; (1) Full-ACT or (2) ACT minus self-as-context (ACT-SAC). Participants in each arm were compared with regards to their ability to engage in psychological flexibility and decentering. Clinical outcomes were compared at end of treatment and also at 6-weeks follow-up.

DETAILED DESCRIPTION:
Acceptance and commitment therapy (ACT) is a 'third wave' behaviour therapy that has been building an evidence base to suggest that it is a promising and useful psychotherapy across a wide range of diagnoses (for reviews see Hayes, Luoma, Bond, Masuda, & Lillis, 2006; Powers, Zum, & Emmelkamp, 2009; Ruiz, 2010; Öst. 2014). ACT is grounded in relational frame theory (RFT; Hayes, 2004) and seeks to define how patients become overly emotionally influenced by internal dialogues, to the point of being immune to positive environmental contingencies (Ciarrochi, Bilich, & Godsel, 2010). The main aim of ACT is to enable psychological flexibility, so that a patient is able to fully connect to the present moment and to also alter (or continue with) behaviours closely aligned to personal values (Hayes et al., 1999). The goal of ACT is to teach skills of handling unwanted/avoided thoughts/feelings to reduce their impact/influence and clarifying what is truly important and meaningful, then using that knowledge to guide, inspire, and motivate continued valued actions in the effort to enrich personal lives (Hayes, 2004).

Psychological flexibility is achieved through six core processes during ACT; defusion; acceptance; contact with the present moment; values; committed action and self-as-context (Hayes, Strosahl, & Wilson, 2012). These components are combined in the 'hexaflex' model (Rolffs, Rogge & Wilson, 2018). Strosahl, Hayes,Wilson, and Gifford (2004) however stated that there was clinically no predefined order for focusing on the processes and not all individuals needed to concentrate on each of the processes to achieve flexibility. There are a variety of in-session and between-session exercises for each aspect of the hexaflex that support patients in understanding, practicing and using the relevant psychological skills (e.g. Hayes et al., 1999).

The ACT model discriminates between three aspects or levels of self; self-as-content, self-as-process, and self-as-context (Hayes et al., 2012). Self-as-content refers to the contents of psychological experience, self-as-process refers to awareness of the on-going changing nature of experiences and self-as-context refers to experiential contact with a persistent and unchanging perspective from which all experiences are observed (De Houwer, Roche, & Dymond, 2013). During ACT, patients learn to build awareness of self-as-context, whilst simultaneously letting go of any over-attachment to a conceptualised self. Self-as-context is independent of content and is the place from which content is observed (Ciarrochi, et al., 2010). The 'I' of self-as-context statements is learnt to be appreciated as stable/constant, in order to retain a sense of self in the face of stress (Pierson et al., 2004) and to appreciate that self-evaluations are transient and temporary (Hayes et al., 1999). Hayes et al (2012) postulated that the ability to occupy a self-as-context position requires self-as-process to be learnt first

The last several decades of psychotherapy outcome research have mainly focussed on gauging the efficacy of 'complete' psychotherapies (i.e. the 'package' of treatment). Whilst this approach has proved useful in some psychotherapies being then recognized as empirically validated, it has simultaneously failed to identify which aspects of the package that are essential, redundant or possibly harmful (Rosen & Davison, 2003). This 'package approach' has also been criticised for promoting the proliferation of apparently 'new' psychotherapies that are essentially re-packages of extant psychotherapies (Ciarrochi et al., 2010). Therefore, despite extensive outcome research validating psychotherapy as an effective treatment (e.g. Roth & Fonagy, 2006), research has been slower to identify the necessary, effective and active ingredients of each individual psychotherapy. Therefore, proving the utility of these different active ingredients (and associated definitive technical features) is a key challenge to the psychotherapy outcome literature (Crits-Christoph, 1997; Stevens, Hynan, & Allen, 2000). Research is therefore necessary that unpacks and compares the components of any psychotherapy 'package' to then assess their relative and specific contribution to outcomes (Stevens et al., 2000).

Two methodological approaches have been previously used to dismantle, isolate and define the importance of specific components within ACT's hexaflex; mediation studies and lab-based component analyses. Mediation analyses index changes in putative processes between treatments, and so identifies the clinical utility of theoretically distinct components (Kraemer, Wilson, Fairburn, & Agras, 2002). However, only a small number of core ACT processes have been examined in mediation studies (namely acceptance and cognitive defusion; see Stockton et al., 2019 for a recent review). Lab-based studies have compared performance on tasks when participants are provided with instructions grounded in a component of the hexaflex (or 'control' instructions) and a meta-analysis has shown small-to-medium effect sizes for 4/6 hexaflex components (Levin, Hildebrandt, Lillis, & Hayes, 2012). No lab-based studies have been conducted on the committed action or self-as-context components (Levin, Hildebrandt, Lillis, & Hayes, 2012). The clinical trial design used to test the efficacy of components of psychotherapies are labelled as either a deconstruction or an additive study (Ahn & Wampold. 2001). Dismantling designs compare a whole treatment, with treatment minus a specific theoretically important component (e.g. Jacobson et al., 1996). Additive designs test the impact of providing a specific and supplementary component hypothesised to enhance outcomes (e.g. Propst, Ostrom, Watkins, Dean, & Mashburn, 1992). No clinical dismantling trials of ACT's hexaflex have been attempted.

RFT provides the theoretical basis for the importance of self-as-context as a component of the hexaflex, as this component is believed to enable and facilitate engagement with the other core processes of the hexaflex (Hayes, 2004). There is however an on-going debate as to whether development of self-as-context is necessary during ACT to enable flexibility, or whether it is sufficient to only develop self-as-process (De Houwer et al., 2013; McHugh & Stewart, 2012). This is the first study to use a deconstruction method to examine the efficacy of the self-as-context component of the psychological flexibility model. Given that the ethical and therapeutic impact of extracting a potentially clinically important hexaflex component has been previously untested, the current study adopted a pilot trial approach. The scientific value of pilot studies that examine the feasibility, safety and effectiveness of new treatments (or in the current context, a deconstructed partial treatment) is widely recognised (Arain, Campbell, Cooper & Lancaster, 2010). The study used participants with a long-term health condition (LTC) and concurrent mental health problems, in terms of their ability to engage in psychological flexibility, decentering and also clinical outcome. Patients with LTCs were seen as an appropriate patient group for the present study, as previous evidence has attested to the effectiveness of ACT with this patient group (Levin et al., 2012). The hypotheses for the study were that participants receiving full ACT would (a) display enhanced ability to engage in psychological flexibility and decentering and (b) achieve better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Long term physical health condition and comorbid mental health problem
* Age 16+
* Referred to a psychological therapies service

Exclusion Criteria:

* Diagnosis of 'medically unexplained symptoms' including somatoform disorders (e.g. pain disorder, conversion disorder, body dysmorphic disorder, hypochondriasis) and functional somatic syndromes (e.g. irritable bowel syndrome, chronic fatigue syndrome, fibromyalgia, non-cardiac chest pain, non-epileptic seizures)
* Mental health diagnoses in addition to anxiety or depression (e.g. personality disorder, bipolar disorder or psychosis)
* Currently accesses secondary care mental health services
* Significant current suicidal risk
* Current substance misuse
* Previous contact with mental health services (defined as two or more prior episodes of service contact without significant change)
* Inpatient admission for mental health difficulties within the last five years
* History of self-injury
* A stated reluctance to engage in psychotherapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Change in psychological flexibility abilities via the Acceptance and Action Questionnaire II (AAQ-II; Bond et al., 2011). | AAQ-II (flexibility) scores compared in the arms at final therapy session and at 6-week follow-up
  The AAQ-II is a 7-item measure of psychological inflexibility (score range 7-49) and is based on the widely researched Acceptance and Action Questionnaire (Hayes et al., 2004). The AAQ-II has sound psychometric properties (Bond et al., 2011).

SECONDARY OUTCOMES:
Change in decentering abilities via the Experiences Questionnaire (EQ; Fresco, Moore, van Dulmen, Segal, Teasdale, Ma, & Williams, 2007). | EQ (decentering) scores compared in the arms at final therapy session and at 6-week follow-up
  The EQ is a 20-item measure of decentering and rumination. Only the EQ-decentering scale was used in the current study; this contains 11-items and so scores ranged from 11-55. The EQ has been shown to have good convergent, discriminant and internal consistency (Fresco, et al., 2007). The EQ-decentering scale has been cross-culturally validated and can detect changes in decentering abilities after mindfulness-based interventions (Soler et al., 2017).

OTHER OUTCOMES:
Change in functioning via the Work and Social Adjustment Scale (WSAS; Mundt, Marks, Shear, & Greist, 2002). | WSAS (functioning) scores compared in the arms at final therapy session and at 6-week follow-up
  The WSAS is a five-item measure of the impact of a health condition on five facets of daily functioning (work, home management, social leisure activities, private leisure activities, and close relationships). All items are scored on a 9-point rating scale from 0 to 8 with a score range of 0-40. Severity ratings are categorised as severe functional impairment >20, significant functional impairment 10-20, subclinical <10). Caseness is defined as scores of ≥10. The WSAS is sensitive to differences in disorder severity and is a sensitive to change (Purdie, Kellett, & Bickerstaffe, 2012).
Changes to depression via The Patient Health Questionnaire (PHQ9; Spitzer, Kroenke & Williams; 1999) | PHQ-9 (depresion) scores compared in the arms at final therapy session and at 6-week follow-up
  The PHQ-9 is a nine-item measure, widely used within primary and secondary care settings to detect depression. All items are scored on a 4-point scale from 0 to 3 with a score range of 0-27. Severity ratings are categorised as severe >20, moderately severe 15-20, moderate 10-14, mild 5-9, remission <5). Caseness is defined as scores of ≥10 and the amount of pre to post treatment change needed to demonstrate statistically reliable change is defined as ≥6 (Gyani, Shafran, Layard, & Clark, 2011). Sensitivity and specificity have been identified at 92% and 80% respectively at the >10 cut off point (Gilbody, Richards, Brealey, & Hewitt, 2007).
Chnages to anxiety via The Generalised Anxiety Disorder Assessment (GAD7; Spitzer, Kroenke, Williams & Lowe; 2006). | GAD-7 (anxiety) scores compared in the arms at final therapy session and at 6-week follow-up
  The GAD-7 is a seven-item severity measure of generalised anxiety. All items are scored on a 4-point scale from 0 to 3 with a score range of 0-21. Severity ratings are categorised as severe >15, moderate 10-14, mild 5-9 & remission <5). Caseness is defined as scores of ≥8 and the amount of pre to post treatment change needed to demonstrate statistically reliable change is defined as ≥4 (Gyani et al., 2011). Applying a threshold score of 10 affords 89% sensitivity and 82% specificity (Swinson, 2006). The GAD-7 has also demonstrated sensitivity and specificity for the detection of other anxiety disorders (e.g. panic disorder, social anxiety disorder; Kroenke, Spitzer, Williams, Monahan & Lowe, 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Thompson, D Clin Psy, Study Director — Director of Research: Clinical Psychology Unit: University of Sheffield
Locations (1):
- Clinical Psychology Unit, Department of Psychology, Uni of Sheffield, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
This will be made apparent in any publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This has been completed
Access Criteria: Other clinical researchers with a validated email address.